CLINICAL TRIAL: NCT02395822
Title: MT2014-25: Haploidentical Donor Natural Killer (NK) Cell Infusion With Subcutaneous Recombinant Human IL-15 (rhIL-15) in Adults With Refractory or Relapsed Acute Myelogenous Leukemia (AML)
Brief Title: MT2014-25: Haplo NK With SQ IL-15 in Adult Relapsed or Refractory AML Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014LS092
Record Dates: First submitted 2015-02-16; First posted 2015-03-24 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2017-12

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Interleukin-15

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preparative Regimen and SubQ rHuIL-15 (Experimental): Preparative Regimen of Fludarabine and Cyclophosphamide
  IL-15 Activation of Donor NK Cells:
  IL-15 to Facilitate NK Cell Survival and Expansion
  Interventions: Biological: IL-15

INTERVENTIONS:
Biological: IL-15 — Preparative Regimen:
  Fludarabine 25 mg/m2 x 5 days start day -6 Cyclophosphamide 60 mg/kg x 2 days on day -5 and -4 (if < 4 months from prior transplant, omit day -4 dose)
  IL-15 Activated Donor NK Cells:
  The apheresis product (collected day -1) will be enriched for NK cells with the large-scale CliniMacs® device (Miltenyi) by depletion of CD3+ cells to remove T-lymphocytes and depletion of CD19+ cells to remove B-lymphocytes. The NK cell enriched product will be activated by overnight incubation with10 ng/ml IL-15 under GMP conditions and infused on day 0.
  IL-15 to Facilitate NK Cell Survival and Expansion:
  IL-15 at 2 mcg/kg subcutaneously (SC) beginning day +1, once a day for 5 days followed by a 2 day rest, and then once a day for 5 days for 10 doses total
  Other Names: Interleukin-15

SUMMARY:
A phase II trial of CD3/CD19 depleted, IL-15 activated, donor natural killer (NK) cells in adults and subcutaneous IL-15 given after a preparative regimen for the treatment of relapsed or refractory acute myelogenous leukemia (AML). The primary objective is to study the potential efficacy of NK cells and IL-15 to achieve complete remission while maintaining safety.

ELIGIBILITY:
Inclusion Criteria (Recipient):

* Meets ONE of the following disease criteria:

  1. Primary AML induction failure: no CR after 2 or more induction attempts
  2. Relapsed AML or Secondary AML (from MDS or treatment related): not in CR after 1 or more cycles of standard re-induction therapy
  3. AML relapsed > 2 months after transplant: No re-induction required, and no more than 1 re-induction cycle is allowed.
  4. Relapsed AML for patients > 60 years of age the 1 cycle of standard chemotherapy is not required if either of the following criteria is met:

     * Relapse within 6 months of last chemotherapy
     * BM blast count < 30% within 10 days of starting protocol therapy
* Available related HLA-haploidentical donor (aged 14 to 75 years) by at least Class I serologic typing at the A&B locus
* Karnofsky Performance Status ≥ 60%
* Patients must have adequate organ within 14 days (28 days for pulmonary and cardiac) of study registration
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to NK cell infusion (excluding preparative regimen pre-medications).
* Agrees to use contraception prior to study entry and for the duration of study participation.

Exclusion Criteria (Recipient):

* Bi-phenotypic acute leukemia.
* Transplant < 60 days prior to study enrollment.
* Active autoimmune disease.
* History of severe asthma
* Uncontrolled intercurrent illness
* New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan that has not been evaluated with bronchoscopy
* Pleural effusion large enough to be detectable on chest x-ray.
* Pregnant women
* History of HIV, active or chronic hepatitis B, hepatitis C or HTLV-I infection
* Known hypersensitivity to any of the study agents used
* Received investigational drugs within the 14 days of study registration.
* Known active CNS involvement.

Criteria For Initial Donor Selection:

* Related donors (sibling, parent, offspring, parent or offspring of an HLA identical sibling).
* 14-75 years of age.
* At least 40 kilogram body weight.
* In general good health as determined by the evaluating medical provider.
* HLA-haploidentical donor/recipient match by at least Class I serologic typing at the A&B locus.
* Not pregnant.
* Able and willing to undergo apheresis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cooley S, He F, Bachanova V, Vercellotti GM, DeFor TE, Curtsinger JM, Robertson P, Grzywacz B, Conlon KC, Waldmann TA, McKenna DH, Blazar BR, Weisdorf DJ, Miller JS. First-in-human trial of rhIL-15 and haploidentical natural killer cell therapy for advanced acute myeloid leukemia. Blood Adv. 2019 Jul 9;3(13):1970-1980. doi: 10.1182/bloodadvances.2018028332. PMID 31266741

RESULTS

PARTICIPANT FLOW:
Groups:
- Preparative Regimen and SubQ rHuIL-15: Preparative Regimen of Fludarabine and Cyclophosphamide
  IL-15 Activation of Donor NK Cells:
  IL-15 to Facilitate NK Cell Survival and Expansion
  IL-15: Preparative Regimen:
  Fludarabine 25 mg/m2 x 5 days start day -6 Cyclophosphamide 60 mg/kg x 2 days on day -5 and -4 (if < 4 months from prior transplant, omit day -4 dose)
  IL-15 Activated Donor NK Cells:
  The apheresis product (collected day -1) will be enriched for NK cells with the large-scale CliniMacs® device (Miltenyi) by depletion of CD3+ cells to remove T-lymphocytes and depletion of CD19+ cells to remove B-lymphocytes. The NK cell enriched product will be activated by overnight incubation with10 ng/ml IL-15 under GMP conditions and infused on day 0.
  IL-15 to Facilitate NK Cell Survival and Expansion:
  IL-15 at 2 mcg/kg subcutaneously (SC) beginning day +1, once a day for 5 days followed by a 2 day rest, and then once a day for 5 days for 10 doses total
Period: Overall Study
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 10
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: < 5% Marrow Blast, no Circulating Peripheral Blasts and Neutrophil Count of > 1 x 10^9/L
Description: Without platelet recovery
Time Frame: Day 42 post NK cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Number analyzed (Participants) | 15
Participants | 5

2. Secondary Outcome: In Vivo Expansion (>100) of NK Cells (Defined at CD56+/CD3- Lymphocytes)
Time Frame: Day 14 post NK cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Number analyzed (Participants) | 15
Participants | 4

3. Secondary Outcome: Proportion of Patients Experiencing Grade, 3, 4, and 5 Toxicities (Assessed by CTCAE v. 4)
Time Frame: Days 1-5 and Days 8-12, 24 hours after the last IL-15 dose, Day +28, Day +42
Measure: Count of Participants; unit: Participants
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Number analyzed (Participants) | 17
Participants | 10

4. Secondary Outcome: Treatment Related Mortality
Time Frame: 6 months post-therapy
Population: 1 patient left the study
Measure: Count of Participants; unit: Participants
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Number analyzed (Participants) | 16
Participants | 2

5. Secondary Outcome: Number of Subjects Achieving Complete Response, Defined as in Vivo Donor Derived NK Cell Expansion of > 100 Donor Derived NK Cells.
Time Frame: Day 42 post NK cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Number analyzed (Participants) | 15
Participants | 1

ADVERSE EVENTS:
Arm/Group | Preparative Regimen and SubQ rHuIL-15
Serious Adverse Events (participants affected / at risk) | 12/17
Other Adverse Events (participants affected / at risk) | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preparative Regimen and SubQ rHuIL-15 (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cytokine Release Syndrome - Grade 3 (Immune system disorders) | 3
Cytokine Release Syndrome - Grade 4 (Immune system disorders) | 2
Abdominal Infection (Infections and infestations) | 1
Endocarditis Infective (Infections and infestations) | 1
Hepatitis Viral (Infections and infestations) | 1
Infections and Infestations - Other, specify (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Intracranial Hemorrhage (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preparative Regimen and SubQ rHuIL-15 (N=17)
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 4
Creatinine increased (Investigations) | 1
Cytokine release syndrome (Immune system disorders) | 5
Encephalopathy (Nervous system disorders) | 2
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 1
Headache (Nervous system disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Weight gain (Investigations) | 5
Mouth/tongue sores (General disorders) | 1
Non Convulsive Status Epilipticus (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No